CLINICAL TRIAL: NCT03489356
Title: Efficacy of a Behavioral Intervention to Reduce Skin Cancer Risk Among Patients
Brief Title: Project Options - The ABC Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kimberly Mallett, Research Associate Professor, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 182279; R21CA196924 (NIH)
Record Dates: First submitted 2018-03-16; First posted 2018-04-05 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Dermatology/Skin - Other; Health Behavior; Sunburn
Keywords: Addressing Behavior Change (ABC); Addressing Behavior Change (ABC) Intervention; Addressing Behavior Change (ABC) Intervention Method
MeSH Terms: conditions — Health Behavior; Sunburn

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Addressing Behavior Change (ABC) intervention delivery method
  Interventions: Behavioral: Addressing Behavior Change (ABC)
- Control (No Intervention): Control

INTERVENTIONS:
Behavioral: Addressing Behavior Change (ABC) — The ABC is a 3-minute brief, dermatologist delivered intervention for dermatological patients that takes place during a skin examination. During the ABC intervention, dermatologists specifically assess patients' UV risk behaviors, discuss patients' motivation to use UV protection, and explore solutions to patient-reported barriers interfering with effective sunscreen use. Based on our previous research, the ABC intervention does not add additional time to the visit, but rather replaces treatment as usual conversations about sun protection.
  Arms: Intervention

SUMMARY:
The present study explores the ability of dermatologists to influence patients' behavior using a novel and brief (3 minute) behavioral intervention in the context of naturally occurring patient interactions and shows promise for long term sustainability. The incidence of invasive skin cancers, cutaneous melanoma in particular, has nearly tripled in the U.S. between 1975 and 2004, making it the fastest rising incidence rate for all cancers in the United States. Dermatologists are in an ideal position to effect change in their patients. The present study will assess whether a brief intervention (The ABC-Addressing Behavior Change method) delivered to patients by dermatologists during a skin examination will increase the use of sun protection and reduce risk behaviors compared to patients who receive treatment as usual.

DETAILED DESCRIPTION:
Skin cancer is the most common malignancy in the U.S. and the incidence and mortality from skin cancer is on the rise. Individuals can decrease their risk of skin cancer by engaging in protective behaviors such as limiting intentional and unintentional UV exposure, and wearing broad-spectrum sunscreens and protective clothing. Despite knowing the risks and receiving dermatological care, many patients with and without a history of skin cancer frequently forget to use UV protection or fail to use it in an optimal manner to reduce their UV risk. To address these concerns, Mallett and colleagues developed a 3-minute brief ABC intervention - Addressing Behavior Change. The ABC intervention is designed to be delivered by dermatologists in the context of a routine office visit involving a skin examination. Previous work by Mallett and colleagues showed dermatologists were highly motivated to deliver the intervention, quickly learned the requisite skills, delivered the intervention with fidelity, and showed minimal decay in knowledge, motivation, and skills over a 6-month period. This study builds on a previous study by conducting an examination of the efficacy of the ABC intervention on patients' motivations and behaviors utilizing a prospective longitudinal design.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for a skin exam with participating dermatologists

Exclusion Criteria:

* psoriasis

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2016-04-25 (Actual); Primary Completion 2017-11-21 (Actual); Study Completion 2017-11-21 (Actual)

PRIMARY OUTCOMES:
Patient Behavior Changes | 1 month and 3 months follow-up
  Examine changes in patients' protective behaviors through surveys; Patients asked for the percent of time they use sunscreen on face, use sunscreen on body, reapply sunscreen often, and cover their skin; Response options range from (0) 0% to (5) 100%

SECONDARY OUTCOMES:
Sunburns | Baseline, 1 month follow-up, 3 month follow-up
  Number of sunburns reported by patients

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly A Mallett, Ph.D., Principal Investigator — Penn State University
Locations (1):
- Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Result] Mallett KA, Turrisi R, Billingsley E, Trager B, Ackerman S, Reavy R, Robinson JK. Evaluation of a Brief Dermatologist-Delivered Intervention vs Usual Care on Sun Protection Behavior. JAMA Dermatol. 2018 Sep 1;154(9):1010-1016. doi: 10.1001/jamadermatol.2018.2331. PMID 30090918

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-23): https://cdn.clinicaltrials.gov/large-docs/56/NCT03489356/Prot_SAP_000.pdf